CLINICAL TRIAL: NCT00508365
Title: A Study to Evaluate the Potential Incidence of Orthostatic Hypotension in Elderly Hypertensive Patients Following Administration of a Combination of COREG CR and Lisinopril
Brief Title: Evaluation of Potential for Orthostatic Hypotension in Elderly Hypertensives
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: CFD109701
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Hypertension
Keywords: lisinopril; carvedilol; hypertension
MeSH Terms: conditions — Hypertension | interventions — Carvedilol; Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects receiving treatment sequence AB (Experimental): Eligible subjects will receive treatment sequence AB; A= Placebo to match COREG CR 20 milligrams once daily plus lisinopril 10 milligrams once daily (Days 1-7). Placebo to match COREG CR 40 milligrams once daily plus lisinopril 10 milligrams once daily (Days 8-14). B=COREG CR 20 milligrams once daily plus lisinopril 10 milligrams once daily (Days 1-7). COREG CR 40 milligrams once daily plus lisinopril 10 milligrams once daily (Days 8-14).
  Interventions: Drug: Carvedilol CR capsules; Drug: Placebo; Drug: Lisinopril
- Subjects receiving treatment sequence BA (Experimental): Eligible subjects will receive treatment sequence BA; B=COREG CR 20 milligrams once daily plus lisinopril 10 milligrams once daily (Days 1-7). COREG CR 40 milligrams once daily plus lisinopril 10 milligrams once daily (Days 8-14). A= Placebo to match COREG CR 20 milligrams once daily plus lisinopril 10 milligrams once daily (Days 1-7). Placebo to match COREG CR 40 milligrams once daily plus lisinopril 10 milligrams once daily (Days 8-14).
  Interventions: Drug: Carvedilol CR capsules; Drug: Placebo; Drug: Lisinopril

INTERVENTIONS:
Drug: Carvedilol CR capsules — The carvedilol micropump (COREG) CR cpsules will be available with doses of 20 milligrams and 40 milligrams administered orally once daily.
Drug: Placebo — Placebo capsules to match each dose level will be provided.
Drug: Lisinopril — Lisinopril will be available as 10 milligrams tablets administered orally once daily.

SUMMARY:
This is a multi-center, double-blind, randomized, placebo-controlled, 2-session crossover study to evaluate the incidence of orthostatic hypotension in elderly hypertensive subjects following co-administration of carvedilol CR and lisinopril.

ELIGIBILITY:
Inclusion Criteria:

* Males or females who are ≥ 65 years of age
* Body mass index (BMI) between 24 and 37 kg/m2 where: BMI = (weight in kg)/ (height in meters)2
* Subjects must have a documented history of essential hypertension and must be stable on treatment with an ACE inhibitor or angiotensin II receptor antagonist or renin antagonist and no more than one other antihypertensive medication at least 3 months before screening with a sitting SBP<180 mmHg and DBP<110 mmHg.
* All subjects must be able to be safely (in the opinion of the Investigator) withdrawn or down-titrated from all antihypertensive treatment(s) and transitioned to lisinopril 10 mg OD for the two-week run-in phase.

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening history, physical or laboratory examination, or any other medical condition or circumstance making the volunteer unsuitable for participation in the study
* Subject who metabolizes carvedilol poorly based on CYP2D6 genotype as determined at screening
* Subject has persistent hyperkalemia or history of hyperkalemia resulting from either Type IV RTA (renal tubular acidosis) or previous treatment with an ACE inhibitor, ARB or renin inhibitor.
* Subject has malignant (accelerated) hypertension, history of malignant hypertension, or history of secondary forms of hypertension
* Subject has advanced hypertensive retinopathy (Keith Wagner Grade IV)
* Subject has a history of hepatic impairment (characterized by prolonged prothrombin time/low concentrations of albumin) and/or renal insufficiency (subjects with an estimated CrCl ≤ 30 mL/min by Cockroft-Gault must be excluded). CrCL = [140-ageCr][weight/70] x 0.85 (if female); Cr in mg/dL; Weight in kg
* Subject is being treated for diabetes mellitus
* Subject has a history of angioedema
* Subject has been under treatment with 3 or more antihypertensive medications. (NOTE: A combination drug containing two antihypertensive agents represents two antihypertensive medications.)
* Subject has been under treatment with HCTZ > 12.5 mg/day
* Subject is receiving ongoing treatment or is anticipated to receive treatment with any of the following medications during the study:

  * monoamine oxidase inhibitors (MAO)
  * any Class I or III antiarrhythmic
  * alpha-adrenergic receptor blockers
  * beta-2-adrenergic agonists
  * all antidepressants including SSRIs
  * lithium
  * medications known to be inhibitors/inducers of cytochrome P-450 2D6 should be discontinued for at least 14 days or 5 half-lives [which ever is longer] prior to the first day of the run-in period
* Treatment with any over-the-counter medications , herbal and dietary supplements, as well as grapefruit-containing products within 7 days or 5 half-lives (whichever is longer) prior to first day of run-in period through the end of the study unless approved by the PI and GSK medical monitor. Standard vitamins and/or daily multi-vitamins are permitted, however herbal vitamins should be excluded.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the run-in period
* Subject has mean sitting SBP ≥ 180 mmHg at the screening assessment (one set of repeat measurement is permitted as per approval by the medical monitor).
* Documented history of low blood pressure within six months of screening visit (average sitting SBP < 110 mm Hg and/or DBP /< 50 mm Hg) or blood pressure below these values at time of screening (one set of repeat measurement is permitted as per approval by the medical monitor).
* Orthostatic hypotension diagnosed at screening (orthostatic hypotension is defined as a reduction in systolic blood pressure of 20 mmHg or more and/or a reduction in diastolic blood pressure of 10 mmHg or more for standing vs. supine measurements)
* Subject has any of the following conditions:

  * uncontrollable or symptomatic arrhythmias; unstable angina
  * sick sinus syndrome or second or third degree heart block (unless treated with a permanent, functioning pacemaker)
  * bradycardia (seated heart rate <55 bpm) (one repeat measurement is permitted as per approval by the medical monitor) ; history of myocardial infarction, or history of stroke within 1 year of screening.
  * subject is in, or has a history of atrial fibrillation
* Any of the following abnormalities on 12-lead ECG during screening:

  * complete RBBB or LBBB
  * evidence of second- or third-degree AV block
  * pathological Q-waves (Q-wave wider than 0.04 sec or depth greater than 0.4-0.5 mV)
  * any other abnormalities that investigator feels could be of concern when patient is taking a β-adrenergic blocking agent
* Donation of blood in excess of 500 mL within a 56-day period including the estimated 150 mL of blood to be drawn during this study
* History of asthma, COPD and/or hypersensitivity to β -adrenergic blocking agents
* History of sensitivity to carvedilol, lisinopril, alpha-blockers, beta-blockers or ACE inhibitors
* History of sensitivity to any of the study medications or components thereof
* History of anaphylaxis or anaphylactoid reactions or severe allergic responses to drugs
* History of regular alcohol consumption exceeding 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening
* Unanticipated positive urine drug screen (UDS) at screening. Note: If the subject is taking a drug known to give a positive on the UDS, then this should be discussed with the medical monitor prior to sending the UDS. In this situation, with prior approval, a positive finding on the UDS will not be considered an exclusion
* Positive for Hepatitis B surface antigen or HIV
* Unwillingness or inability to follow the procedures outlined in the protocol or inability to provide written informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-09-25 (Actual); Primary Completion 2008-06-03 (Actual); Study Completion 2008-06-03 (Actual)

PRIMARY OUTCOMES:
Assessment of orthostasis 6 hours post dose on day 1, 7, 8, 14 in each dosing session | 6 hours post dose on day 1, 7, 8, 14 in each dosing session
To evaluate the incidence of orthostatic hypotension (defined as a decrease in SBP of ≥20 mmHg and/or a decrease in DBP of ≥10 mmHg in changing from the supine to the standing position) following co-administration of COREG CR and lisinopril | Up to Day 14

SECONDARY OUTCOMES:
Relationship of concentration of drug to events 6 hours post dose on day 1, 7, 8, 14 in each dosing session | 6 hours post dose on day 1, 7, 8, 14 in each dosing session
Relationship of concentration of drug to events | 6 hours post dose on day 1, 7, 8, 14 in each dosing session
To evaluate the safety and tolerability of the co-administration of COREG CR and lisinopril | Up to Day 24
To evaluate the relationship between the plasma concentrations of carvedilol and lisinopril and the occurrence of orthostatic hypotension following co-administration of COREG CR and lisinopril | 6 hours post dose on day 1, 7, 8, 14 in each dosing session
To evaluate the effects of COREG CR on plasma renin activity | Up to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- United States (20):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] GSK has submitted manuscripts of these study results to peer-reviewed scientific journals which were not accepted for publication. GSK is providing the attached study results summary with a conclusion.
- See also: Results for study CFD109701 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/CFD109701?search=study&study_ids=CFD109701#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: CFD109701 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: CFD109701 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: CFD109701 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: CFD109701 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: CFD109701 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: CFD109701 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: CFD109701 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register